CLINICAL TRIAL: NCT02139904
Title: A Randomised Phase II Trial of Oral Vinorelbine as Second Line Therapy for Patients With Malignant Pleural Mesothelioma
Brief Title: Vinorelbine in Mesothelioma
Acronym: VIM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wales Cancer Trials Unit (Other)
Collaborators: Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UNOLE 0329
Record Dates: First submitted 2014-05-09; First posted 2014-05-15 (Estimated); Last update posted 2021-10-12 (Actual); Status verified 2021-10

CONDITIONS: Mesothelioma
Keywords: Mesothelioma; Vinorelbine; BRCA1
MeSH Terms: conditions — Mesothelioma | interventions — Vinorelbine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Symptom Control (Placebo Comparator): Active symptom control includes palliative care and standard care methods used to manage symptoms
  Interventions: Other: Active Symptom Control
- Vinorelbine (Active Comparator): Active symptom control (ASC) as per local practice plus vinorelbine administered at a dose of 60mg/m2 orally on day 1, day 8 and day 15 on a 3- weekly cycle, incrementing to 80mg/m2 weekly on a 3-weekly cycle in the absence of any significant toxicity for subsequent cycles. Patients will continue chemotherapy until evidence of radiological progression (or unacceptable toxicity or patient withdrawal).
  Interventions: Drug: Vinorelbine

INTERVENTIONS:
Drug: Vinorelbine — Vinorelbine was first licensed in the UK for Non-Small Cell Lung Cancer (NSCLC) and advanced breast cancer in 1997. Vinorelbine (Navelbine®) is a semi-synthetic, third generation, vinca alkaloid. The cytotoxic effect of vinorelbine is through the disruption of mitotic spindle formation, blocking mitosis at the G2-M stage resulting in cell death.
  Other Names: Navelbine
  Arms: Vinorelbine
Other: Active Symptom Control
  Arms: Active Symptom Control

SUMMARY:
This study is for patients with malignant mesothelioma of the lung lining (called pleura) who have had previous chemotherapy with a platinum-based regimen whose disease has progressed. Malignant pleural mesothelioma (MPM) is an aggressive, frequently drug resistant, and incurable disease that is increasing in incidence in the UK and worldwide. All patients with MPM will relapse following first line chemotherapy and at present, there is no standard treatment available for patients in the second line setting. The vinca alkaloid chemotherapy drug vinorelbine has shown promising activity in a single arm UK trial. However to date, there has been no randomised evaluation of vinorelbine in mesothelioma in the second line setting. In addition, there have been no trials which have looked at underlying molecular changes in mesothelioma which may predict vinorelbine efficacy; This might allow vinorelbine to be used in patients only where there is a chance of benefit. Studies suggest that vinorelbine requires a gene called BRCA1 (shown to be absent in 38% of mesothelioma cases) in order to induce cell death in mesothelioma. The VIM trial aims to establish whether vinorelbine in patients with MPM helps them live longer and whether the BRCA1 gene is helpful in selecting patients most likely to benefit from treatment.

Patients will be randomised (1:2) to receive either active symptom control (ASC) (which is all supportive care deemed necessary for pain management excluding disease modifying treatment) or ASC with vinorelbine. Patients will continue vinorelbine treatment until evidence of disease progression (or unacceptable toxicity to the drug or patient withdrawal). If vinorelbine activity is demonstrated, we will use the results from this trial to inform the design of a future phase III trial.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed histological diagnosis of malignant pleural mesothelioma. The same block or 10 unstained slides should be available for translational research
2. Prior treatment with first-line standard platinum doublet based chemotherapy only
3. Evidence of disease progression according to CT scan
4. Life expectancy ≥ 3 months
5. ECOG performance status 0-2
6. Men or women aged 18 years or over
7. Willing to consent to provide blood and tissue for translational research
8. Measurable lesions by modified RECIST
9. Adequate organ function, including the following: Adequate bone marrow reserve: absolute neutrophil count (ANC) ≥ 1.5 x 109/L, WBC >3 x 109/L, haemoglobin ≥ 100g/L, platelets ≥ 100 x 109/L; adequate liver function: Bilirubin <1.5 x ULN AST/ALT 1.5- 2.5 x ULN.
10. Patients with reproductive potential (male or female), who are sexually active during the duration of the trial or the drug washout period, should be prepared to use two effective forms of contraception throughout their participation in the trial and for at least three months after the last dose of vinorelbine.
11. Patients must provide informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Patients with a diagnosis of a second malignancy except prostate or cervical cancer in remission or patients with a diagnosis of basal cell carcinoma of the skin.
2. Have received treatment with an agent that has not received regulatory approval, within 30 days of study entry.
3. Are pregnant or breastfeeding.
4. Uncontrolled CNS disease.
5. Known contraindication or hypersensitivity to vinorelbine or other vinca alkaloids or to any of the constituents
6. Any disease significantly affecting absorption
7. Previous significant surgical resection of stomach or small bowel
8. Yellow fever vaccine within 30 days of consent
9. Previous vinca alkaloid chemotherapy
10. Palliative radiotherapy within the RECIST area in the 4 weeks prior to baseline CT chest up until randomisation.
11. Patients that are unable to swallow

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2021-03-17 (Actual); Study Completion 2021-03-17 (Actual)

PRIMARY OUTCOMES:
Overall Survival | 2 years
  Anti-tumour activity of vinorelbine will be measured by overall survival, time from randomisation to death.

SECONDARY OUTCOMES:
Progression Free Survival | 2 years
  Anti-tumour activity of vinorelbine will also be measured by progression free survival. We will document time from randomisation to any disease progression and/or death, defined according to strict RECIST v1.1. Lesions will be compared with baseline measurements to assess progression
Number of serious adverse events reported | 2 years
  The toxicity profile of oral vinorelbine in this setting will be used to assess safety. An independent data monitoring committee will convene and assess safety 6 months after the first patient has been randomised. If the trial is deemed safe to continue then safety will be assessed again approx every 6 months. Toxicity data will be assessed alongside serious adverse events.
BRCA1 status in blood and tumour samples | 2 years
  Tumour and blood samples will be collected for future translational research. BRCA1 expression as a putative predictor of vinorelbine sensitivity will be measured primarily in the samples.

CONTACTS AND LOCATIONS:
Overall Officials: Dean Fennell, Professor, Study Chair — University of Leicester
Locations (1):
- Wales Cancer Trials Unit, Cardiff, United Kingdom

REFERENCES:
- [Derived] Fennell DA, Porter C, Lester J, Danson S, Taylor P, Sheaff M, Rudd RM, Gaba A, Busacca S, Nixon L, Gardner G, Darlison L, Poile C, Richards C, Jordan PW, Griffiths G, Casbard A. Active symptom control with or without oral vinorelbine in patients with relapsed malignant pleural mesothelioma (VIM): A randomised, phase 2 trial. EClinicalMedicine. 2022 May 19;48:101432. doi: 10.1016/j.eclinm.2022.101432. eCollection 2022 Jun. PMID 35706488
- See also: Related trial information — https://www.cardiff.ac.uk/centre-for-trials-research